CLINICAL TRIAL: NCT06269367
Title: NewGait: A Low-Cost Rehabilitation System to Improve Post-Stroke Gait (Biomechanical Adaptations)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Chandramouli Krishnan, Associate Professor of Physical Medicine and Rehabilitation, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HUM00226149; 1R41HD111289-01 (NIH)
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: gait training; balance; Stroke survivors
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the two device interventions but will receive both interventions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NewGait (Experimental): Participants will put on the NewGait device and walk on the treadmill and overground. Participants may receive biofeedback of their gait patterns to engage them in the training.
  Interventions: Other: NewGait
- Control (Other): Participants will put on the Control device and walk on the treadmill and over ground. Participants may receive biofeedback of their gait patterns to engage them in the training.
  Interventions: Other: Control wearable limb orthotic device

INTERVENTIONS:
Other: NewGait — wearable limb orthotic device
  Arms: NewGait
Other: Control wearable limb orthotic device — wearable limb orthotic device
  Arms: Control

SUMMARY:
An affordable and easy to use gait-assistive device for stroke survivors to use at home is yet to be developed. This study is intended to modify the current design of the NewGait device to specifically work for stroke survivors based on feedback from patients and clinicians. Consequently, conducting a short-term biomechanical gait study is planned to determine the usability and functionality of the NewGait device compared to other comparative devices.

DETAILED DESCRIPTION:
More than 795,000 individuals suffer from a stroke each year in the United States, making stroke a leading cause of adult disability in the United States and worldwide. More than half of stroke survivors exhibit reduced independence and functional mobility due to stroke-related gait impairments. Despite significant advancements in post-stroke medical care and rehabilitation, current treatments are not successful in optimally restoring gait function after stroke. It is well established that intense, repetitive task-oriented rehabilitation interventions are essential for inducing experience-dependent neuroplasticity (defined as the ability of the nervous system to adapt and optimize its resources through structural and functional changes)-which is a key factor for post-stroke gait recovery. Accordingly, new therapeutic approaches that rely on specialized gait training devices, such as treadmills, robotic devices, and exosuits have been developed. However, these devices are typically expensive, bulky, and not accessible for home use. Moreover, these devices often require uninterrupted power sources, which is a major barrier for rural communities in developing nations. While some lightweight and "low-cost" commercial devices exist, they are not often designed based on multi-user feedback and robust biomechanical data and their clinical utility have not been tested in stroke survivors, thereby limiting usability and effectiveness. Thus, there is a significant unmet clinical need for an effective, affordable, and portable gait mobility/rehabilitation device that is accessible for most stroke survivors. This Phase-I STTR pursues the following specific aims: (1) Identify an optimal NewGait design based on end-user feedback (design sprints) and musculoskeletal modeling to address the needs of stroke rehabilitation, (2) Refine the current prototype using data gathered from design sprints and think aloud technique and perform benchtop testing on the final prototype to validate durability, and (3) Examine short-term gait adaptations and clinical feasibility in stroke survivors by performing a comparative clinical feasibility study in stroke survivors to establish the clinical utility of the NewGait device in comparison with other similar devices. This trial registration is for the third aim only, as the first two aims do not follow under the definition of clinical trial. All devices tested are deemed to be 501(k) exempt devices. The successful completion of this Phase-I STTR will lay the foundation for an evidence-based low-cost gait rehabilitation system that could positively affect the lives of millions of stroke survivors living across the globe.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral cortical or subcortical stroke
* Chronic stroke (≥ 6 months) At least 6 months following their first unilateral stroke
* Able to walk independently with/without assistive devices for 5-10 mins (~150m)
* No significant cognitive deficits as determined by the Mini Mental State Examination (MMSE) score (score≥ 22)

Exclusion Criteria:

* Cerebellar stroke
* Traumatic or vascular brain injury
* History of unstable heart condition, uncontrolled diabetes/hypertension
* History of a recent lower-extremity trauma or fracture
* History of a recent significant orthopedic or neurological conditions that could limit walking ability (e.g., multiple sclerosis, total knee replacement)
* Documented history of significant spatial neglect
* ankle joint contractures or significant spasticity in the lower limbs
* History of a recent Botulinum Toxin (Botox) injection to the lower-extremity muscles (≤ 3 months)
* Pregnant or actively planning to become pregnant (self-reported)- Inability to communicate or unable to consent

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandramouli Krishnan, PT, PhD, Principal Investigator — University of Michigan
Locations (1):
- Physical Medicine & Rehabilitation 325 E Eisenhower Pkwy Suite 3011, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NewGait/Control: Participants will put on the NewGait device and walk on the treadmill and overground. Participants may receive biofeedback of their gait patterns to engage them in the training.
  NewGait: wearable limb orthotic device
  Following this, participants will put on the Control device and walk on the treadmill and overground. Participants may receive biofeedback of their gait patterns to engage them in the training.
  Control wearable limb orthotic device: wearable limb orthotic device
- Control/NewGait: Participants will put on the Control device and walk on the treadmill and overground. Participants may receive biofeedback of their gait patterns to engage them in the training.
  Control wearable limb orthotic device: wearable limb orthotic device
  Following this, participants will put on the NewGait device and walk on the treadmill and overground. Participants may receive biofeedback of their gait patterns to engage them in the training.
  NewGait: wearable limb orthotic device
Period: Phase I
Arm/Group | NewGait/Control | Control/NewGait
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Not completed — Unable to perform study procedures | 0 | 1
Not completed — Could not continue study for personal reasons. | 1 | 0
Period: Phase II
Arm/Group | NewGait/Control | Control/NewGait
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NewGait/Control | Control/NewGait | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (7.8) | 64.6 (7.2) | 64.1 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 4 | 8 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 9 | 6 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Mini-mental state examination score [Mean (Standard Deviation); unit: units on a scale] — Measure of cognitive function on a scale of 0 to 30, with higher scores representing greater cognitive function.
  units on a scale | 28.9 (1.9) | 28.0 (1.9) | 28.5 (1.9)
Time since stroke [Mean (Standard Deviation); unit: months] | 102.3 (47.8) | 136.2 (94.9) | 119.3 (75.2)
Lower extremity Fugl-Meyer score [Mean (Standard Deviation); unit: units on a scale] — Measure of lower extremity impairment post-stroke on a scale from 0 to 34, with a higher score representing less impairment.
  units on a scale | 21.8 (3.4) | 22.3 (4.3) | 22.1 (3.8)
Gait speed [Mean (Standard Deviation); unit: meters per second] — Measure of preferred walking speed from 0 to no upper limit, with a higher value indicating faster walking speed.
  meters per second | 0.9 (0.4) | 0.9 (0.3) | 0.9 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Gait Speed
Description: Changes in gait speed (from baseline) as measured using the 10 Meter Walk Test between the experimental (NewGait) and control conditions. Participants were timed during the 10 Meter Walk Test to determine their self-selected gait speed while walking overground in a hallway. In this test, participants walked down a 14 meter walkway, and a stopwatch was used to time how long it took participants to cross the intermediate 10 meter distance. The baseline measure for the first device was taken immediately prior to the intervention. Participants then wore the first device, and the during-training measure was taken immediately. After this, participants received training with the device for about 15 minutes, following which, the device was removed and the post-intervention measure was taken immediately for the first device. Participants then rested for 20-30 minutes. This entire process was repeated with the second device. All measures were obtained on the same day.
Time Frame: Up to 2 hours
Population: Data was only analyzed on participants who completed the study.
Measure: Mean (Standard Error); unit: meters per second
Arm/Group | NewGait | Control
Number analyzed (Participants) | 18 | 18
meters per second
  Baseline | 0.90 (0.09) | 0.92 (0.08)
  During training | 0.88 (0.08) | 0.87 (0.08)
  Post-intervention | 0.91 (0.09) | 0.92 (0.09)
Statistical Analysis 1: Comparison: NewGait vs Control; Test type: Superiority; p = 0.894, ANOVA; Two way repeated measures ANOVA with time (Baseline, post-intervention) and condition (NewGait, Control) as within-subjects factors

2. Primary Outcome: Ankle Muscle Activation
Description: Changes in ankle muscle activation of the leg muscles as measured using surface electromyography between the experimental (NewGait) and control conditions. Muscle activation ranges from 0 to no upper limit, and higher activation meant that the muscle was being used more. The baseline measure for the first device was taken immediately prior to the intervention. Participants then wore the first device, and the during-training measure was taken immediately. After this, participants received training with the device for about 15 minutes, following which, the device was removed, and the post-intervention measure was taken immediately for the first device. Participants then rested for 20-30 minutes. This entire process was repeated with the second device. All measures were obtained on the same day.
Time Frame: Up to 2 hours
Population: Data was only analyzed on participants who completed the study.
Measure: Mean (Standard Error); unit: percentage of maximum muscle activation
Arm/Group | NewGait | Control
Number analyzed (Participants) | 18 | 18
percentage of maximum muscle activation
  Medial Gastrocnemius, Baseline | 75.29 (15.68) | 72.98 (15.68)
  Medial Gastrocnemius, During training | 62.41 (14.61) | 66.77 (15.05)
  Medial Gastrocnemius, Post-intervention | 67.77 (15.26) | 75.46 (15.12)
  Lateral Soleus, Baseline | 68.61 (14.78) | 68.43 (14.41)
  Lateral Soleus, During training | 72.72 (14.22) | 72.24 (13.49)
  Lateral Soleus, Post-intervention | 68.66 (15.99) | 64.05 (15.99)
  Tibialis Anterior, Baseline | 30.87 (2.93) | 30.08 (3.83)
  Tibialis Anterior, During training | 28.04 (3.87) | 21.55 (3.87)
  Tibialis Anterior, Post-intervention | 25.71 (4.04) | 30.02 (3.02)
Statistical Analysis 1: Comparison: NewGait vs Control; Test type: Superiority; p > 0.299, ANOVA — A priori threshold for statistical significance was set to 0.05; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Changes in Paretic Leg Propulsive Force
Description: Changes in paretic leg propulsive force were measured using ground reaction forces obtained from force sensors during walking between the experimental (NewGait) and control conditions. Propulsive force had no upper or lower limit, with a higher number indicating greater propulsion from the paretic limb. The baseline measure for the first device was taken immediately prior to the intervention. Participants then wore the first device, and the during-training measure was taken immediately. After this, participants received training with the device for about 15 minutes, following which, the device was removed, and the post-intervention measure was taken immediately for the first device. Participants then rested for 20-30 minutes. This entire process was repeated with the second device. Results reflect Newton units in force generated divided by Newton units of body weight (N/N) times 100. All measures were obtained on the same day.
Time Frame: Up to 2 hours
Population: Data was only analyzed on participants who completed the study.
Measure: Mean (Standard Error); unit: percentage of body weight (N/N)
Arm/Group | NewGait | Control
Number analyzed (Participants) | 18 | 18
percentage of body weight (N/N)
  Baseline | 8.22 (1.26) | 8.03 (1.26)
  During training | 11.92 (1.86) | 11.36 (1.86)
  Post-intervention | 8.70 (1.31) | 9.00 (1.31)
Statistical Analysis 1: Comparison: NewGait vs Control; Test type: Superiority; p = 0.469, ANOVA — A priori threshold for statistical significance set to 0.05; [statistical method as in outcome 1, analysis 1]

4. Other Pre Specified Outcome: Changes in Paretic Leg Loading (i.e., Vertical Ground Reaction Force)
Description: Changes in paretic leg loading were measured using vertical ground reaction forces obtained from force sensors during walking between the experimental (NewGait) and control conditions.
Time Frame: Up to 2 hours
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Changes in Other Lower Extremity Muscle Activation
Description: Changes in lower extremity muscle activation as measured using surface electromyography between the experimental (NewGait) and control conditions.
Time Frame: Up to 2 hours
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Muscle Coordination
Description: Changes in ankle muscle coordination of the leg muscles as measured using surface electromyography between the experimental (NewGait) and control conditions.
Time Frame: Up to 2 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 hours
Arm/Group | NewGait | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 14/20 | 14/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NewGait (N=20) | Control (N=20)
Skin Irritation (Skin and subcutaneous tissue disorders) | 4 | 4
Muscle/Joint Pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Fatigue (Musculoskeletal and connective tissue disorders) | 9 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT06269367/Prot_SAP_001.pdf
  • Informed Consent Form (2024-11-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT06269367/ICF_000.pdf